CLINICAL TRIAL: NCT03029273
Title: Pilot Study of Affinity-enhanced Anti-NY-ESO-1 TCR Engineered Autologous T Cells in NSCLC Patients
Brief Title: NY-ESO-1 TCR （TAEST16001）for Patients With Advanced NSCLC
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangzhou Institute of Respiratory Disease (Other)
Collaborators: Xiangxue Life Science Research Center (Unknown); Guangdong Xiangxue Precision Medical Technology Co., Ltd. (Industry); Xiangxue Pharmaceutical (Other)
Responsible Party: Principal Investigator, ShiYue Li, MD,Professor, Guangzhou Institute of Respiratory Disease
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-63
Record Dates: First submitted 2017-01-20; First posted 2017-01-24 (Estimated); Last update posted 2019-01-17 (Actual); Status verified 2019-01

CONDITIONS: Lung Cancer, Nonsmall Cell, Recurrent
MeSH Terms: conditions — Lung Neoplasms; Recurrence | interventions — Cyclophosphamide; fludarabine

STUDY DESIGN:
Intervention Model Description: One arm, open label, dose escalation, single dose phase I study of safety and tolerability.
  NYESO-1 TCR-T cell are prepared via lentiviral infection. DLT was administered in a dose escalation test according to the 3 + 3 design. Seven days prior to infusion of TCR-T cell, subjects receive cytoreductive chemotherapy with cyclophosphamide (250-500mg/m2/day) plus fludarabine (25mg/m2/day) for 3 days.
  Patients, who receive an infusion of TAEST16001, will remain in the hospital to be monitored for adverse events until they have recovered from the treatment.
  Patients will have frequent follow-up visit to monitor the persistence of modified T cells and efficacy of the treatment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anti-NY-ESO-1 TCR-transduced T cells (Experimental): NYESO-1 TCR-T cell are prepared via lentiviral infection. DLT was administered in a dose escalation test according to the 3 + 3 design. Seven days prior to infusion of TCR-T cell, subjects receive cytoreductive chemotherapy with Cyclophosphamide (250-500mg/m2/day) and Fludarabine (25mg/m2/day) for 3 days.
  A single dose of Anti-NY-ESO-1 TCR transduced T cells (about 5×109) will be intravenously (i.v.) administered Additionally, following infusion of Anti-NY-ESO-1 TCR transduced T cells, IL-2 subcutaneous injections (500,000 IU/day) will be administered for 14 days concomitantly to each subject.
  Interventions: Drug: Cyclophosphamide and Fludarabine; Biological: Anti-NY-ESO-1 TCR transduced T cells

INTERVENTIONS:
Drug: Cyclophosphamide and Fludarabine — Seven days prior to infusion of TCR-T cell, subjects receive cytoreductive chemotherapy with cyclophosphamide (250-500mg/m2/day) plus fludarabine (25mg/m2/day) for 3 days.
Biological: Anti-NY-ESO-1 TCR transduced T cells — A single dose of Anti-NY-ESO-1 TCR transduced T cells (about 5×109) will be intravenously (i.v.) administered Additionally, following infusion of Anti-NY-ESO-1 TCR transduced T cells, IL-2 subcutaneous injections (500,000 IU/day) will be administered for 14 days concomitantly to each subject.

SUMMARY:
TCR-T cell therapy experienced a breakthrough for treating tumors in recent years. Phase I / II trial of NY-ESO-1-specific TCR-T treatment for synovial sarcoma and melanoma conducted by the Rosenberg team at the National Cancer Institute showed that 61% Synovial cell sarcoma and 55% melanoma had therapeutic responses. Another report of a phase I / II clinical trial for multiple myeloma showed that 20 patients received high affinity anti-NY-ESO-1 and LAGE-1 specific TCR-T treatment, 16 of them (80%) had the average progression-free survival of 19.1 months with minor side effect. These achievements indicate that TCR-T cell therapy can target a variety of tumors including solid tumors without any severe side effects found in CAR-T trials.

This study is mainly focused on tumor testis antigen (Cancer-Testis Antigen), because it is not expressed in normal cells. NY-ESO-1 antigen is commonly expressed in 10-50% of melanoma, lung, liver, esophageal, breast, prostate, bladder, thyroid and ovarian cancer cases, 60% of multiple myeloma cases, and 70-80% of synovial cell sarcoma. Approximately 700,000 new cases of lung cancer are identified each year in China, 70% of them die within one to two years after diagnosis due to the lack of effective treatment. To address that unmet needs, our TCR-T treatment targets non-small cell lung cancer with NY-ESO-1 antigen expression.

This study will investigate the safety and tolerability of TAEST16001 (TAEST: TCR Affinity Enhancing Specific T cell Therapy, autologous T cells transduced with affinity enhanced NY-ESO-1 TCR) cell therapy in subjects with NSCLC who have received prior therapy for their disease but their disease has progressed or relapsed.

DETAILED DESCRIPTION:
This Phase 1 study is designed as a cell dose escalation trial evaluating the safety of TAEST16001 T cell therapy in subjects with NSCLC who have received prior therapy for their disease but the disease has progressed or relapsed. Anti-tumor activity and other exploratory objectives will be assessed. Subjects enter from a Screening Protocol and are positive for HLA-A2*02:01 and have tumor that express NY-ESO-1. The subjects will be evaluated DLT and MTD using a modified 3+3 cell dose escalation design to determine the cell dose range. Subjects will receive cytoreductive chemotherapy with cyclophosphamide (250-500mg/m2/day) plus fludarabine (25mg/m2/day) on day -7 to day -5 followed by infusion of dose of about 5×109 TAEST16001 and IL-2(s.c.).

Subjects will stay in hospital for safety and efficacy assessment daily from T cell infusion (Day 0) through Day 7, and then weekly until week 4 and then at 8 weeks, 12 weeks, 16 weeks and every 3 months until progression of their disease.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 and ≤75 years old while signing the informed consent;
2. Sign an informed consent before undertaking any trial-related activities;
3. Stage IIIb-IV NSCLC patients diagnosed by licensed pathologist, NY-ESO-1 positive cells >10% by IHC.
4. Received at least one run of standard therapy(surgery, chemo, radiation and targeted therapy) or first line and second line treatment failure; If the patient has EGFR mutation or ALK gene rearrangement, they can be enrolled after the appropriate EGFR or ALK tyrosine kinase inhibitor treatment failed;
5. Have one positive indication of the following immunological biomarkers during the screening stage: HLA-A*0201+, NYESO-1+;
6. ECOG score 0-1(see appendix);Life expectancy is longer than 3 months;
7. No Chinese herbal medicine usage within 4 weeks before enrollment;
8. left ventricular ejection fraction≥50%
9. Lab test results meet the following requirements:

   White blood cell count≥3.0×109/L; ANC≥1.5 ×109/L (No GCSF support); PLT≥75 ×109/L; Hemoglobin≥10g/dL (No transfusion in the last 7 days); Prothrombin time or INR ≤1.5× normal upper limit, except taking anticoagulant therapy; PTT≤1.5× normal upper limit, except taking Anticoagulant therapy;a 24-hour creatinine clearance rate≥60mL/ min; AST/SGOT≤2.5 ×ULN; ALT/SGPT≤2.5 ×ULN; ALP≤2.5 ×ULN; TBIL≤1.5×ULN (expect that the subject has Gilber's syndrome).
10. Levels of calcium, potassium, and magnesium in serum are within the normal range;
11. Pregnancy test is negative for female subjects with reproductive capability before participating the study；Female subjects must consent using birth control during the study or prohibit any homo or heterosexual behavior;
12. Can regularly visit the research institutions for tests, evaluations, and monitoring throughout the study period.

Exclusion Criteria:

1. SCLC;
2. Received major surgery, conventional chemotherapy, large-area radiotherapy, immune therapy or any biological anti-tumor therapy within 4 weeks prior to the study;
3. Allergic to any components of the therapy;
4. Never recovered to <2 grade CTCAE from prior surgery or treatment-related adverse events;
5. With two types of primary solid tumors;
6. Poorly managed hypertension (systolic blood pressure >160 mmHg and / or diastolic blood pressure > 90 mmHg) or clinically significant(for example, active) cardiovascular and cerebrovascular diseases such as cerebrovascular incident (within 6 months prior to signing the informed consent), myocardial infarction (within 6 months prior to signing the informed consent), unstable angina, grade II or above heart failure according to New York Heart Association Grading (See Appendix) Congestive, or severe arrhythmia can not be controlled by medication or has a potential impact on the study; With consecutive three times of obvious abnormality on electrocardiogram or average QTc interval ≥450 ms;
7. With other serious organic disease and/or mental illness;
8. With systemic active infections that need treatments, including active tuberculosis, HIV-positive or clinically active hepatitis A, B and C;
9. With autoimmune diseases: such as a history of inflammatory bowel disease (IBD) or other autoimmune diseases determined by the investigator to be unsuitable for the study (e.g. systemic lupus erythematosus (SLE), vasculitis, invasive pulmonary disease);
10. Within 4 weeks prior the infusion, received chronic systemic steroid cortisone, Hydroxyurea, immunomodulatory treatment (for example: Interleukin 2, alpha or gamma interferon, GCSF, mTOR inhibitors, cyclosporine etc.);
11. History of organ allografts, autologous / allogeneic stem cell transplantation, and renal replacement therapy;
12. With central nervous system metastasis. Patients with neurological symptoms need a brain CT/MRI examination to rule out brain metastases;
13. With uncontrolled diabetes, pulmonary fibrosis, interstitial lung disease, acute lung disease, or liver failure;
14. History of alcohol and / or drug abuse;
15. Pregnant or lactating female patients;
16. Received concomitant medication prohibited by the protocol;
17. With any medical condition or disease determined by the investigators that may be detrimental to this trial;
18. No capacity or limited capacity to make juridical acts.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-03-21 (Actual); Primary Completion 2019-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events | 30 Days
  To evaluate the safety and feasibility of the administration of anti-NY-ESO-1 TCR transduced T cells in patients with HLA-A2+ NY-ESO-1 expressing NSCLC.

SECONDARY OUTCOMES:
Number of participants with clinical responses | 270 Days
  To evaluate the efficacy of NYESO-1 positive NSCLS patients treated with NY-ESO-1 antigen specific affinity-enhanced TCR transduced autologous T cell therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Shiyue Li, MD, Principal Investigator — Guangzhou Institute of Respiratory Disease, The First Affiliated Hospital of Guangzhou Medical University; Chengzhi Zhou, MD, Principal Investigator — Guangzhou Institute of Respiratory Disease, The First Affiliated Hospital of Guangzhou Medical University
Locations (1):
- Guangzhou Institute of Respiratory Disease, The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided